CLINICAL TRIAL: NCT05780489
Title: Evaluation of Salivary ELISA for Hormone Monitoring in Donors
Acronym: MINT-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Collaborators: MINT DIAGNOSTICS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2211-VLC-158-EB
Record Dates: First submitted 2023-02-28; First posted 2023-03-22 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Infertility, Female; Reproductive Sterility
Keywords: SALIVA; DONNORS; OESTRADIOL; PROGESTERONE
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Intervention Model Description: This is a prospective multicentric study,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DONORS UNDER CONTROLLED OVARIAN STIMULATION (Experimental): Saliva samples will be analyzed using oestradiol and progesterone ELISA kits.
  Interventions: Diagnostic Test: Determination of progesterone and oestradiol

INTERVENTIONS:
Diagnostic Test: Determination of progesterone and oestradiol — Blood and saliva samples will be taken for determination of progesterone and oestradiol hormones.

SUMMARY:
In donors or patients undergoing assisted reproduction treatments (ART) it is necessary to closely control ovarian stimulation to monitor the number and size of developing follicles.

Oestradiol (E2) and progesterone (P4) are products of steroidogenesis. Their concentrations increase with the diameter of the growing follicle. In order to assess treatment response and support clinical decisions, accurate and reliable methods to measure E2 and P4 are essential. Measurement of both hormones, as well as monitoring of follicle growth through ultrasound measurements, is an important part of ovarian stimulation, requiring patients or donors to undergo multiple blood draws. It is often a physically and emotionally painful process, and the most convenient solution is the measurement of hormones concentrations in other biological fluids, such as saliva. Salivary diagnostic tests are a less invasive, inexpensive, and stress-free alternative.

The current study pretends to evaluate the correlation between salivary ELISA assays and serum determination of progesterone and oestradiol concentrations in oocyte donors, and, also, evaluate the feasibility of doing saliva E2 and P4 determinations in the IVIRMA clinic labs.

ELIGIBILITY:
Inclusion criteria

* Informed consent form dated and signed
* Woman undergoing COS for oocyte donation
* Age 18-35, inclusive
* Regular menstrual cycles
* In good health and not suffering from any mental or medical condition(s) that would preclude participation in the study

Exclusion criteria

• Simultaneous participation in other clinical study, that at the investigator's criteria could interfere with the results of this study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
E2 and P4 on Day 1 | 1 YEAR
  Measurement of saliva E2 adn P4 values on day 1 stimulation
E2 and P4 on Day 8 | 1 YEAR
  Measurement of saliva E2 adn P4 values on day 8 of stimulation
E2 and P4 on Triggering day | 1 YEAR
  Measurement of saliva E2 adn P4 values on triggering day

SECONDARY OUTCOMES:
BODY MASS INDEX | 1 year
  Measurement of body mass index
DONOR'S AGE | 1 year
  Age at the procedure moment
NUMBER OF OOCYTES | 1 YEAR
  Number of oocytes collected

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Ivi Madrid, Madrid
  - IVI Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No